CLINICAL TRIAL: NCT05332600
Title: Assessment Protocol on Lower Limbs Aligment Pre and Post Muscular Fatigue During DROP-JUMP TEST
Brief Title: Pre and Post Muscular Fatigue - DROP-JUMP TEST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculdade de Ciências Médicas da Santa Casa de São Paulo (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: DROP-JUMP TEST
Record Dates: First submitted 2022-02-09; First posted 2022-04-18 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Motor Control
Keywords: rehabilitation; lower limb-muscle; alignment, sequence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pre and post fatigue assessment (Experimental): assessment pre and post fatigue protocol
  Interventions: Other: drop-jump test

INTERVENTIONS:
Other: drop-jump test — The participants will be submitted to a kinematic evaluation protocol before and after fatigue protocol and after two weeks they will be submitted again to the same protocol, however, they will be guided and trained on the correct execution of the tested movement.

SUMMARY:
Many studies have related the presence of dynamic valgus with several musculoskeletal injuries of the hip, knee and ankle. The weakness of the hip abductors is cited as one of the factors linked to this poor dynamic alignment of the lower limb, however, motor control can also be one of the factors responsible for the poor alignment of the lower limbs.

ELIGIBILITY:
Inclusion Criteria:

Women aged between 18 and 29 years body mass index between 18.5 and 24.99 sedentary irregularly active no pain no injuries (hip, knee, foot, ankle or lumbar spine) no neurological sequelae

Exclusion Criteria:

pain during the test

Ages: 18 Years to 29 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — female, 18 years (minimum) and 29 years (maximum)
Enrollment: 35 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
lower limb motor control | assessment pre fatigue
  pre fatigue - DROP-JUMP test
lower limb motor control | assessment pos fatigue up to 01 week
  post fatigue - DROP-JUMP test

CONTACTS AND LOCATIONS:
Locations (1):
- ISCMSP, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided